CLINICAL TRIAL: NCT01874600
Title: A Pivotal, Phase III Trial of Detecting Generalized Tonic-Clonic Seizures With a Seizure Detection and Warning System in Epilepsy Patients
Brief Title: Seizure Detection and Warning System for Epilepsy Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brain Sentinel (Other)
Responsible Party: Sponsor
Other Study IDs: BS-0421
Record Dates: First submitted 2013-06-05; First posted 2013-06-11 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epilepsy Patients: This study will compare accuracy of seizure detection by the study device to simultaneously collected data of seizure detection by video EEG.
  Interventions: Device: Brain Sentinel Seizure Detection Device and Warning System

INTERVENTIONS:
Device: Brain Sentinel Seizure Detection Device and Warning System — The Brain Sentinel Seizure Detection Device and Warning System is designed to monitor Epilepsy patients and alerts caregivers that a GTC seizure is occurring

SUMMARY:
The seizure detection and warning system is an ambulatory system designed to monitor and analyze EMG data to detect the onset of GTC seizures and to provide a warning signal to alert caregivers that a seizure is occurring.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a suspected history of GTC seizures, either primary GTC or partial onset seizures with secondary generalization.
2. Is being admitted to a hospital for routine vEEG monitoring related to seizures.
3. Male or female between the ages of 13-21.
4. If female and of childbearing potential, has a negative pregnancy urine test, and must also not be nursing.
5. Can understand and sign written informed consent, or will have a parent or a legally authorized representative (LAR) who can do so, prior to the performance of any study assessments.
6. Subject and/or Primary Caregiver must be competent to follow all study procedures.
7. Is able to read, speak, and understand English or has a LAR that does so.
8. Subject/LAR consents to the use of vEEG files, including video/audio recordings, for purposes of this research study.

Exclusion Criteria:

1. Has not had a GTC seizure within the last year AND is not expected to have a reduction of anti-epileptic drugs during their hospital admission.
2. Intracranial EEG electrodes are being used.
3. The subject is allergic to adhesives or any component of the electrode patch assembly

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent epilepsy patients with a history of generalized tonic-clonic seizures either primary GTC or partial onset seizures with second generalization.
Sampling Method: Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2013-07; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome is accuracy of device to detect GTC seizures when compared to video EEG. | less than 1 month
  The primary objective of the research is to determine the ability of the Brain Sentinel Seizure Detection System to accurately detect GTC seizures in comparison to the recognized "gold standard" for seizure detection, video Electroencephalography (vEEG).The primary endpoint will be the sensitivity of GTC seizure detection (defined as within 30 seconds of motor manifestation via vEEG analysis) in a hospital setting.

SECONDARY OUTCOMES:
Comparison of study device to self reporting of seizures using a seizure diary. | Less than 1 month
  The secondary objective is to assess the operation of the Brain Sentinel Seizure Detection System when used in the subject's home and to compare the GTC seizure reporting of the device to a standard seizure diary completed by the subject/caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Jose' E Cavazos, MD, PhD, Principal Investigator — Brain Sentinel; Dennis Dlugos, MD, Principal Investigator — Children's Hospital of Philadelphia; Jonathan Halford, MD, Principal Investigator — Medical University of South Carolina; Dileep Nair, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Brain Sentinel, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No